CLINICAL TRIAL: NCT02238015
Title: To Investigate Tear Film Change After Phacoemulsification With SS-OCT
Brief Title: Tear Film Evaluation After Phacoemulsification
Acronym: TFAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zheng Qian (Other)
Responsible Party: Sponsor-Investigator, Zheng Qian, Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: WZMC2013BNZYJ
Record Dates: First submitted 2014-08-28; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Cortical Senile Cataract
Keywords: cataract ,tear film,SS-OCT
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- surgery group: patients underwent cataract surgery with 3.0 mm clear corneal incision at 11 o'clock in one eye
  Interventions: Procedure: cataract surgery
- control group: patients' other eye that did not have surgery

INTERVENTIONS:
Procedure: cataract surgery — All patients underwent cataract surgery with 3.0 mm clear corneal incision at 11 o'clock in one eye
  Groups: surgery group

SUMMARY:
To compare tear film differences between surgical eyes and nonsurgical eyes in patients who had cataract surgery by phacoemulsification in one eye.

DETAILED DESCRIPTION:
All participants granted their written informed consent to participate in the research protocol.

ELIGIBILITY:
Inclusion Criteria:

age-related cataract without surgery history and dry eye symptoms history

Exclusion Criteria:

diseases influencing tear secretion (such as Sjögren syndrome, Steve-Johnson syndrome, diabetes, thyroid disease, etc.); history of ocular surgeries or nuclear hardness IV and V, which required the use of larger phacoemulsification energy; use of drugs that affect tear secretion and stability (such as glaucoma medications, artificial tears, corticosteroid drugs, etc.); or presence of ocular diseases (such as Pterygium, blepharitis, uveitis, glaucoma, lacrimal apparatus, etc.).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 eyes from 30 age-related cataract participants underwent cataract surgery with 3.0 mm clear corneal incision at 11 o'clock in one eye and the other eye without surgery history
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Phacoemulsification influence on the postoperative tear functions | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qian Zheng, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China